CLINICAL TRIAL: NCT02591693
Title: Feasibility Study: Improving Caregiver Confidence in Their Ability to Look After Patients With Palliative Care Needs, Using Focused One to One Training in the Home
Brief Title: Individualised Informal Caregiver Training for Palliative Care at Home
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial OT left post due to significant personal circumstances. Study team unable to recruit new OT to post in time frame available.
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other); Oxford Brookes University (Other); University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REC number 14/SC/1104
Record Dates: First submitted 2015-09-29; First posted 2015-10-29 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Palliative Care
Keywords: Family Caregivers; Occupational Therapy; Activities of Daily Living

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caregiver Training (Experimental): Three home visits by a specialist occupational therapist, each lasting 1-2 hours. Assessment and training to confidently achieve up to three goals relating to practical activities of daily living identified by patient and caregiver.
  On-going usual care from multi-professional team at hospice.
  Interventions: Behavioral: Caregiver training
- Usual Care (No Intervention): On-going usual care from multi-professional team at hospice.

INTERVENTIONS:
Behavioral: Caregiver training — Occupational therapy training focuses on improving confidence to manage practical aspects of care in areas of daily life important to patient and caregiver, in which caregiver reports or anticipates low levels of confidence.
  Arms: Caregiver Training

SUMMARY:
The purpose of this study is to determine whether a training intervention to improve caregiver confidence for family caregivers of patients with palliative care needs at home, is acceptable to patients and their caregivers.

DETAILED DESCRIPTION:
Many patients with terminal illnesses rely on friends and family for much of their practical day to day care. These friends and family members often lack the skills and confidence to carry out these tasks and studies have shown that many would want more support. Studies have also shown that many patients feel they are a burden.

This study involves carers receiving training to learn the skills they need to care for their loved one. Adult patients with terminal illnesses, currently receiving care from a specified hospice in the South East of England, who have a friend or family member caring for them at home are eligible to be referred for this study.

The training of the carer will be carried out over three sessions by an Occupational Therapist in the patient's own home.The training will focus on goals that the patient and carer have chosen together.

The carer will be asked to complete before and after questionnaires and some will be asked to take part in interviews to see how they felt about the study.

The potential benefits of this study are to increase carer confidence in caring for their loved one.

The overall aim of this study is to test out the research method to see if patients and carers find this training and the outcome measures acceptable. If they do then the investigators plan to learn from this study to design a larger randomised control trial which would be the best way of knowing for sure whether and in what ways this training is helpful.

ELIGIBILITY:
Inclusion Criteria:

* Patient currently at home, reliant on family/friends (lay carers) some or all of the time to help with practical or personal care.
* The carer is aged 18 years or over.
* The carer and the patient have the capacity to consent to being involved in the study.

Exclusion Criteria:

* There is a current plan in place for all care to be provided by paid carers full time.
* The patient currently receiving more than one contact with Hospice Specialist Occupational Therapy or is likely to develop needs requiring more than one contact Hospice Occupational Therapy over the four week study intervention period.
* Patients and carers who are not able to speak or understand adequate English for consent to be obtained, to be able to undertake carer training and to complete the study outcome measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Recruitment, retention, attrition, missing data rates | 6 weeks post recruitment
  To evaluate feasibility of study

SECONDARY OUTCOMES:
Preparedness for caregiving scale | Baseline and 4-6 weeks
  Validated for carers of patients with dementia but is used in palliative care settings. Eight items evaluate carer preparedness to care across multiple domains of caregiving. Items rated on a 5 point scale. Low scores indicate less preparedness.
Caregiver Burden Scale at End of Life | Baseline and 4-6 weeks
  Validated for use in carers looking after patients with chronic illness. 14 items measured on a 5 point scale evaluate perceived difficulty in completing tasks. High scores indicate greater burden.
Modified Caregiver Strain Index | Baseline and 4-6 weeks
  13 item tool developed for carers looking after older adults living in community based settings. Items measure strain related to care provision in financial, physical, psychological, social or personal domains scored on a three point scale. High scores indicate higher levels of strain.
Carer Confidence Scale | Baseline and 4-6 weeks
  Non validated. Developed by research team as no existing tools measure carer confidence in palliative care settings. A single question asks carers to rate their confidence to care on a 5 point scale. Higher scores indicate greater confidence.

OTHER OUTCOMES:
Health care utilisation | 4-6 weeks
  A record of unplanned or emergency care accessed by patient over course of study period will be completed by carers.
Acceptability | 4-6 weeks
  Carer and patient questionnaires, carer qualitative interviews, occupational therapist report
Age | Baseline
  Patient and carer demographics will be collected.
Gender | Baseline
Diagnosis | Baseline
  Diagnosis of patient
Health status | Baseline
  Self reported health status of carer
Co-morbidities | Baseline
  Other medical conditions
Social Circumstances | Baseline
  Lives alone, lives with, type of housing,

CONTACTS AND LOCATIONS:
Overall Officials: Bee Wee, MB BCh PhD, Study Chair — Oxford University Hospitals NHS Trust and University of Oxford
Locations (1):
- Sir Michael Sobell House Hospice, Oxford, Oxfordshire, United Kingdom